CLINICAL TRIAL: NCT03008655
Title: A Split-face Comparison of Low Fluence 1064-nm Q-switched Nd:YAG Laser Plus Vitamin C vs Low Fluence 1064-nm Q-switched Nd:YAG Laser Plus Intradermal Tranexamic Acid Injection for Melasma:a Single Blinded, Randomised Study
Brief Title: 1064-nm Q-switched Nd:YAG Laser and Intradermal Tranexamic Acid for Melasma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Principal Investigator, Huang Yu Chen, Attending physician of Dermatology Department, Taipei Medical University WanFang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N201610008
Record Dates: First submitted 2016-12-22; First posted 2017-01-02 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-12

CONDITIONS: Melasma
MeSH Terms: conditions — Melanosis | interventions — Lasers, Solid-State

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nd-YAG (Active Comparator): ND-YAG only
  Interventions: Device: Nd-YAG
- Nd-YAG and intradermal tranexamic acid (Experimental): Nd-YAG combine with intradermal tranexamic acid
  Interventions: Procedure: intradermal tranexamic acid; Device: Nd-YAG

INTERVENTIONS:
Procedure: intradermal tranexamic acid — intradermal tranexamic acid injection
  Arms: Nd-YAG and intradermal tranexamic acid
Device: Nd-YAG — six session at two-week interval of low influence 1064 Nd:YAG laser (6 mm spot size, energy fluence 1.2 - 1.4 J/cm 2 at 10 Hz)

SUMMARY:
BACKGROUND: Melasma is a chronic, often relapsing skin disorder, with poor long-term results from all current therapies.Q switched 1064nm Nd:YAG laser and intradermal tranexamic acid both showed efficacy on the treatment of melasma. However, no combination therapy of both be reported.

OBJECTIVES: To compare the efficacy of low influence Q switched 1064nm Nd:YAG laser and low influence Q switched 1064nm Nd:YAG laser combined with intradermal tranexamic acid injection for melasma.

DETAILED DESCRIPTION:
METHODS: Twenty patients with melasma were included in a randomized controlled observer-blinded study with split-face design. Each side of the face was randomly allocated to either six session at two-week interval of low influence 1064 Nd:YAG laser (6 mm spot size, energy fluence 1.2 - 1.4 J/cm 2 at 10 Hz) or low influence 1064nm Nd:YAG laser combined with intradermal tranexamic acid injection.Complication Improvement of melasma was assessed by Melasma area severity index (MASI),physician's global assessment (PhGA), MELASQOL scale, patient's global assessment (PGA), and patient's satisfaction at baseline,6th week,10th week after first treatment and 3 months, and 6 months after last treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients > 20 years old with refractory melasma to topical treatment

Exclusion Criteria:

* History of keloid, active eczema, active acne in the face, history of facial eczema, photosensitivity, use of isotretinoin in the past 6 months, pregnancy, and high exposure to sunlight or UV light (UVA or UVB)

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Melasma area severity index (MASI) | 6 months after last treatment

SECONDARY OUTCOMES:
Quality of life by MELASQOL scale | 6th week,10th week after first treatment and 3 months, and 6 months after last treatment
Improvement by patient's global assessment (PGA), | 6th week,10th week after first treatment and 3 months, and 6 months after last treatment
Patient's satisfaction (VAS) | 6th week,10th week after first treatment and 3 months, and 6 months after last treatment
Improvement by physician's global assessment (PhGA) | 6th week,10th week after first treatment and 3 months, and 6 months after last treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yu Chen Huang, MD, Principal Investigator — Taipei Medical University WanFang Hospital

IPD SHARING:
Plan to Share IPD: No